CLINICAL TRIAL: NCT00354133
Title: The Effect of Deep Brain Stimulation of the Subthalamic Nucleus (STN-DBS) on Quality of Life in Comparison to Best Medical Treatment in Patients With Complicated Parkinson's Disease and Preserved Psychosocial Competence (EARLYSTIM-study)
Brief Title: Controlled Trial With Deep Brain Stimulation in Patients With Early Parkinson's Disease
Acronym: EARLYSTIM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Parkinson Study Group (GPS) (Other)
Collaborators: University Hospital Schleswig-Holstein (Other); Assistance Publique - Hôpitaux de Paris (Other); KKS Netzwerk (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A 121/06
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Deep Brain Stimulation; PDQ-39
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBS treatment (Active Comparator): Patients in this arm are treated with Deep Brain Stimulation (DBS) of the Nucleus subthalamicus with the device Kinetra and Soletra (neurostimulator, Medtronic) and addtionally get best medical treatment
  Interventions: Device: Kinetra and Soletra (neurostimulator, Medtronic)
- BMT treatment (Active Comparator): Patients in this arm get best medical treatment only.
  Interventions: Drug: Best Medical Treatment

INTERVENTIONS:
Device: Kinetra and Soletra (neurostimulator, Medtronic) — Patients in this arm were implanted with a neurostimulator (Kinetra and Soletra from Medtronic) are stimulated. Additionally the get best medical treatment.
  Arms: DBS treatment
Drug: Best Medical Treatment — Patients in this arm get best medical treatment only
  Arms: BMT treatment

SUMMARY:
Earlystim Study: Patients are randomized either to medical treatment or subthalamic stimulation. The observation period was 2 years. The primary outcome criterium: PDQ-39.

Post study Follow up studies: After the 24 months observation period also BMT patients could be operated and all patients will be observed for 10 years or longer to elucidate whether earlier stimulation has advantages (or drawbacks) compared to later stimulation.

DETAILED DESCRIPTION:
Parkinsons' disease is one of the most disabling chronic neurological diseases. It can be treated sufficiently until motor complications with fluctuations of mobility and dyskinesias develop. The quality of life and the social and occupational functioning is relentlessly deteriorating with longer disease duration once the complications of conservative therapy develop. High-frequency stimulation of the subthalamic nucleus especially improves the motor complications of Parkinson's disease and preliminary data suggest that also the quality of life and psychosocial handicap are improved. So far this therapy is only used for patients which have already undergone personal, professional and social degradation due to motor complications of the disease. The aim of this study is to assess the use of this therapy in earlier stages of the disease, when motor complications have just developed and before patients are significantly affected in their social and occupational functioning.

The main study (Earlystim) was finished in March 2012 and published in February 2013 (Schuepbach WM, Rau J, Knudsen K, et al. Neurostimulation for Parkinson's disease with early motor complications. N Engl J Med. Feb 14 2013;368(7):610-622.) Patients, who were treated with BMT only in the Earlystim Study were privileged to be operated after the 24 months and a follow up phase of 5 years was planned to elucidate whether earlier stimulation has advantages (or drawbacks) compared to later stimulation.

As operated patients fare better in terms of quality of life and other outcomes (see publication), it will be important to know if patients who are operated earlier keep an advantage in all thoses parameters over those who were operated later or if those operated later will catch up after surgery. Also the pattern of adverse events among earlier and later operated patients may differ. These issues can be addressed with the post-study follow-up (PSFU) studies of the patients of the Earlystim trial. The results of these investigations elucidate longterm issues of DBS in PD and may affect the recommendations of surgery for patients.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease
* Hoehn and Yahr stage ≤ 2.5 in the best "on"med condition
* Disease duration > 4 years
* Presence of fluctuations and/or dyskinesias for no more than 3 years
* One of the two following forms of impairment:
* Impairment in activities of daily living (UPDRS II > 6) due to PD-symptoms despite medical treatment in the "worst" condition or
* Impairment of social and occupational functioning (measured with a modified SOFAS) due to PD-symptoms despite medical treatment (51-80%)
* PDQ-39 completed
* Written informed consent
* For the patients in France a social security number is required

Exclusion Criteria

* Major depression with suicidal thoughts (Beck Depression Inventory > 25)
* Dementia (Mattis Score ≤ 130)
* Acute psychosis
* Need for nursing care
* Any medical or psychological problems which may interfere with a smooth conduction of the study protocol (e.g. cancer with a limited life expectancy)
* Drug or alcohol addiction
* Surgical contraindications
* Fertile women not using adequate contraceptive methods
* Women who are pregnant or breast feeding
* Illiteracy or insufficient language skills (German or French) to complete the questionnaires
* Simultaneous participation in another clinical trial except that other trial does not affect the Earlystim study as approved and documented by the steering committee

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2006-07; Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
PDQ-39 | 24 months
  Difference in the PDQ-39 summary index at 24 months compared to the baseline assessment.

SECONDARY OUTCOMES:
UPDRS part III | 24 months
  Change in the Unified Parkinson's disease Rating Scale (UPDRS) part III
UPDRS II scale | 24 months
  Change in the UPDRS II scale
Safety | 24 months
  Frequency, type and severity of therapy related adverse events of medication or DBS, Change in medication (L-DOPA equivalents)
UPDRS VI scale | 24 months
  Change in the UPDRS VI scale
SCOPA-PS | 24 months
  Change in the SCOPA-PS scale
BDI scale | 24 months
  Change in the BDI scale
MADRS scale | 24 months
  Change in the MADRS scale
BPRS scale | 24 months
  Change in the BPRS scale
Mattis Dementia Scale | 24 months
  Change in the Mattis Dementia Scale
Ardouin Behaviour Scale | 24 months
  Change in the Ardouin Behaviour Scale
Starkstein-Apathy Scale | 24 months
  Change in the Starkstein-Apathy Scale
professional Fitness scale | 24 months
  Change in the professional Fitness scale
SF-36 scale | 24 months
  Change in the SF-36 scale
pain (VAS) scale, | 24 months
  Change in the pain (VAS) scale
clinical global impression (CGI-GI) scale | 24 months
  change in the clinical global impression (CGI-GI) scale
"best"-state | 24 months
  Change in the number of hours per day in the "best"-state
"best" state dyskinesias | 24 months
  Frequency and severity of "best" state dyskinesias
Sleeping-hours per day | 24 months
  Sleeping-hours per day
Gait | 24 months
  Changes in gait
Speech | 24 months
  Changes in speech

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Deuschl, Prof., Principal Investigator — Department of Neurology, Christian-Albrechts-University Kiel, Schittenhelmstr. 10, D 24105 Kiel; Marie Vidailhet, Prof., Principal Investigator — Groupe Hospitalier Pitié- Salpêtrière, Fédération des Maladies du Système Nerveux, 47-83 Boulevard de l´Hôpital, F- 75651 Paris Cedex 13
Locations (16):
- France (8):
  - Michallon Hospital, CHU Grenoble, Service de Neurologie, BP217, Grenoble
  - Service de Neurologie C, Hôpital Neurologique et neurochirurgical Pierre Wertheimer , 59 Bd Pinel 69677 BRON Cedex, Lyon
  - Centre hospitalier La Timone, Service de neurologie et pathologie du mouvement,Boulevard Jean Moulin, Marseille
  - "Hôpital Nord Laënnec Boulevard Jacques-Monod - Saint-Herblain, Nantes
  - CIC, CHU Pitié-Salpêtrière, 47-83 Bd de l'Hôpital, Paris
  - Hôpital La Milétrie, Tour Jean Bernard, 350 Av Jacques Cœur, BP 577, Poitiers
  - Centre Hospitalo-Universitaire de Rouen, Charles Nicolle, bat. DV, 1 rue de Germont, Rouen
  - Centre d'investigation Clinique, Pavillon Riser, Hôpital Purpan,Place du Dr Baylac TSA 40031, Toulouse
- Germany (8):
  - Klinik und Poliklinik für Neurologie, Charite, Berlin
  - Klinik und Poliklinik für Neurologie, Cologne
  - Neurologische Klinik der Universität, Moorenstr. 5, Düsseldorf
  - Neurologische Universitätsklinik Freiburg, Breisacher Str. 64, Freiburg im Breisgau
  - Paracelsus-Elena-Klinik, Kassel, Klinikstrasse 16, Kassel
  - Klinik für Neurologie, Universitätsklinikum Schleswig-Holstein, Schittenhelmstr. 10, Kiel
  - Klinikum der Universität München Neurologische Klinik und Poliklinik - Großhadern, Marchioninistr. 15, München
  - Universitätsklinikum Tübingen, Klinik für Neurochirurgie, Hoppe-Seyler-Str.3, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: by inidividual contact with the Coordinatin Investigator Prof.Dr. Deuschl

REFERENCES:
- [Result] Schuepbach WM, Rau J, Knudsen K, Volkmann J, Krack P, Timmermann L, Halbig TD, Hesekamp H, Navarro SM, Meier N, Falk D, Mehdorn M, Paschen S, Maarouf M, Barbe MT, Fink GR, Kupsch A, Gruber D, Schneider GH, Seigneuret E, Kistner A, Chaynes P, Ory-Magne F, Brefel Courbon C, Vesper J, Schnitzler A, Wojtecki L, Houeto JL, Bataille B, Maltete D, Damier P, Raoul S, Sixel-Doering F, Hellwig D, Gharabaghi A, Kruger R, Pinsker MO, Amtage F, Regis JM, Witjas T, Thobois S, Mertens P, Kloss M, Hartmann A, Oertel WH, Post B, Speelman H, Agid Y, Schade-Brittinger C, Deuschl G; EARLYSTIM Study Group. Neurostimulation for Parkinson's disease with early motor complications. N Engl J Med. 2013 Feb 14;368(7):610-22. doi: 10.1056/NEJMoa1205158. PMID 23406026
- [Result] Deuschl G, Schade-Brittinger C, Agid Y; EARLYSTIM Study Group. Neurostimulation for Parkinson's disease with early motor complications. N Engl J Med. 2013 May 23;368(21):2038. doi: 10.1056/NEJMc1303485. No abstract available. PMID 23697520
- [Result] Dams J, Balzer-Geldsetzer M, Siebert U, Deuschl G, Schuepbach WM, Krack P, Timmermann L, Schnitzler A, Reese JP, Dodel R; EARLYSTIM-investigators. Cost-effectiveness of neurostimulation in Parkinson's disease with early motor complications. Mov Disord. 2016 Aug;31(8):1183-91. doi: 10.1002/mds.26740. PMID 27506638
- [Result] Lhommee E, Wojtecki L, Czernecki V, Witt K, Maier F, Tonder L, Timmermann L, Halbig TD, Pineau F, Durif F, Witjas T, Pinsker M, Mehdorn M, Sixel-Doring F, Kupsch A, Kruger R, Elben S, Chabardes S, Thobois S, Brefel-Courbon C, Ory-Magne F, Regis JM, Maltete D, Sauvaget A, Rau J, Schnitzler A, Schupbach M, Schade-Brittinger C, Deuschl G, Houeto JL, Krack P; EARLYSTIM study group. Behavioural outcomes of subthalamic stimulation and medical therapy versus medical therapy alone for Parkinson's disease with early motor complications (EARLYSTIM trial): secondary analysis of an open-label randomised trial. Lancet Neurol. 2018 Mar;17(3):223-231. doi: 10.1016/S1474-4422(18)30035-8. PMID 29452685
- [Result] Schupbach WM, Rau J, Houeto JL, Krack P, Schnitzler A, Schade-Brittinger C, Timmermann L, Deuschl G. Myths and facts about the EARLYSTIM study. Mov Disord. 2014 Dec;29(14):1742-50. doi: 10.1002/mds.26080. Epub 2014 Nov 14. PMID 25399678
- [Result] Deuschl G, Schupbach M, Knudsen K, Pinsker MO, Cornu P, Rau J, Agid Y, Schade-Brittinger C. Stimulation of the subthalamic nucleus at an earlier disease stage of Parkinson's disease: concept and standards of the EARLYSTIM-study. Parkinsonism Relat Disord. 2013 Jan;19(1):56-61. doi: 10.1016/j.parkreldis.2012.07.004. Epub 2012 Jul 28. PMID 22841616
- [Derived] Pinto S, Nebel A, Rau J, Espesser R, Maillochon P, Niebuhr O, Krack P, Witjas T, Ghio A, Cuartero MC, Timmermann L, Schnitzler A, Hesekamp H, Meier N, Mullner J, Halbig TD, Moller B, Paschen S, Paschen L, Volkmann J, Barbe MT, Fink GR, Becker J, Reker P, Kuhn AA, Schneider GH, Fraix V, Seigneuret E, Kistner A, Rascol O, Brefel-Courbon C, Ory-Magne F, Hartmann CJ, Wojtecki L, Fradet A, Maltete D, Damier P, Le Dily S, Sixel-Doring F, Benecke P, Weiss D, Wachter T, Pinsker MO, Regis J, Thobois S, Polo G, Houeto JL, Hartmann A, Knudsen K, Vidailhet M, Schupbach M, Deuschl G; EARLYSTIM Study Group. Results of a Randomized Clinical Trial of Speech After Early Neurostimulation in Parkinson's Disease. Mov Disord. 2023 Feb;38(2):212-222. doi: 10.1002/mds.29282. Epub 2022 Dec 3. PMID 36461899
- [Derived] Schuepbach WMM, Tonder L, Schnitzler A, Krack P, Rau J, Hartmann A, Halbig TD, Pineau F, Falk A, Paschen L, Paschen S, Volkmann J, Dafsari HS, Barbe MT, Fink GR, Kuhn A, Kupsch A, Schneider GH, Seigneuret E, Fraix V, Kistner A, Chaynes PP, Ory-Magne F, Brefel-Courbon C, Vesper J, Wojtecki L, Derrey S, Maltete D, Damier P, Derkinderen P, Sixel-Doring F, Trenkwalder C, Gharabaghi A, Wachter T, Weiss D, Pinsker MO, Regis JM, Witjas T, Thobois S, Mertens P, Knudsen K, Schade-Brittinger C, Houeto JL, Agid Y, Vidailhet M, Timmermann L, Deuschl G; EARLYSTIM study group. Quality of life predicts outcome of deep brain stimulation in early Parkinson disease. Neurology. 2019 Mar 5;92(10):e1109-e1120. doi: 10.1212/WNL.0000000000007037. Epub 2019 Feb 8. PMID 30737338
- See also: (German Research Collaboration, funded by the German Ministry of Research) — http://www.kompetenznetz-parkinson.de/
- See also: (Homepage Coordination Center for Clinical Studies to STN Study, Language: German) — http://www.kks.uni-marburg.de/
- See also: Schuepbach WM, Rau J, Knudsen K, et al. Neurostimulation for Parkinson's disease with early motor complications. N Engl J Med. Feb 14 2013;368(7):610-622. — http://www.kks.uni-marburg.de/